CLINICAL TRIAL: NCT00127205
Title: Phase III Trial of Bisphosphonates as Adjuvant Therapy for Primary Breast Cancer
Brief Title: S0307 Phase III Trial of Bisphosphonates as Adjuvant Therapy for Primary Breast Cancer.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); North Central Cancer Treatment Group (Network); Eastern Cooperative Oncology Group (Network); NSABP Foundation Inc (Network); Cancer and Leukemia Group B (Network); NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000437061; S0307 (Other: SWOG)
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Clodronic Acid; Ibandronic Acid; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (Experimental): Patients receive zoledronate IV over 15 minutes once a month for 6 months and then once every 3 months for 2.5 years.
  Interventions: Drug: zoledronic acid
- Arm II (Active Comparator): Patients receive oral clodronate once daily for 35 months.
  Interventions: Drug: clodronate disodium
- Arm III (Experimental): Patients receive oral ibandronate once daily for 35 months.
  Interventions: Drug: ibandronate sodium

INTERVENTIONS:
Drug: clodronate disodium — Given orally
  Arms: Arm II
Drug: ibandronate sodium — Given orally
  Arms: Arm III
Drug: zoledronic acid — Given IV
  Arms: Arm I

SUMMARY:
RATIONALE: Zoledronate, clodronate, or ibandronate may delay or prevent bone metastases in patients with nonmetastatic breast cancer. It is not yet known whether zoledronate is more effective than clodronate or ibandronate in treating breast cancer.

PURPOSE: This randomized phase III trial is studying zoledronate to see how well it works compared to clodronate or ibandronate in treating women who have undergone surgery for stage I, stage II, or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare disease-free survival and overall survival of women with resected primary stage I-III adenocarcinoma of the breast treated with adjuvant zoledronate vs clodronate vs ibandronate.
* Compare the distributions of sites of first disease recurrence in patients treated with these drugs.
* Compare adverse events in patients treated with these drugs.
* Correlate parathyroid hormone related protein status and N-telopeptide levels at baseline with disease-free survival and sites of first recurrence in patients treated with these drugs.
* Investigate whether there is an association between inherited germ-line single nucleotide polymorphisms (SNP, rs2297480) in farnesyl diphosphate synthase (FDPS) and the adverse event of acute phase reactions in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive zoledronate IV over 15 minutes once a month for 6 months and then once every 3 months for 2.5 years.
* Arm II: Patients receive oral clodronate once daily for 35 months.
* Arm III: Patients receive oral ibandronate once daily for 35 months. Treatment in all arms continues in the absence of disease recurrence or unacceptable toxicity.

After completion of study treatment, patients are followed every 6 months until disease recurrence and then annually for up to 10 years.

PROJECTED ACCRUAL: A total of 5,400 will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary adenocarcinoma of the breast

  * Stage I-III disease
  * No evidence of metastatic disease
* Must have undergone lumpectomy or total mastectomy for primary disease within the past 12 weeks, or have completed chemotherapy within the past 8 weeks

  * Axillary evaluation per institutional standards
* Currently receiving or planning to receive standard adjuvant systemic therapy comprising chemotherapy, hormonal therapy, or combined chemotherapy/hormonal therapy for breast cancer

  * Patients who are at low risk for disease recurrence and for whom adjuvant systemic therapy will not be prescribed are not eligible
  * Patients who receive biologic agents only or local radiotherapy only (without chemotherapy and/or hormone therapy) are not eligible
  * Additional therapies are allowed including radiotherapy and biologic agents (e.g., trastuzumab [Herceptin^®], bevacizumab, or hematopoietic growth factors)
  * Neoadjuvant therapy or hormonal therapy alone is allowed provided study entry occurs ≥ 12 weeks after completion of surgery
* Patients with skeletal pain are eligible provided bone scan and/or roentgenological exam are negative for metastatic disease

  * Suspicious findings must be confirmed as benign by x-ray, MRI, or biopsy
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Creatinine ≤ 2 times upper limit of normal
* Creatinine clearance ≥ 30 mL/min
* No renal failure

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of esophageal stricture or motility disorders

  * Gastroesophageal reflux disorder allowed
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior or concurrent hematopoietic growth factors allowed
* HER-2-targeted therapies allowed
* Antiangiogenics allowed

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* Concurrent radiotherapy to the breast, chest wall, or lymph node group allowed at the discretion of the treating physician

Surgery

* See Disease Characteristics

Other

* Prior neoadjuvant therapy allowed
* Prior bisphosphonates for bone density allowed
* No other concurrent bisphosphonates as adjuvant therapy or for treatment of osteoporosis
* No concurrent enrollment in clinical trials with bone density as an endpoint

  * Concurrent enrollment on any other locoregional or systemic therapy breast cancer study (including cooperative group studies) allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6097 (Actual)
Dates: Start 2005-07; Primary Completion 2017-12 (Actual); Study Completion 2021-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie R. Gralow, MD, Study Chair — Seattle Cancer Care Alliance; Robert B. Livingston, MD, Study Chair — University of Arizona; James N. Ingle, MD, Study Chair — Mayo Clinic; Carla I. Falkson, MD, Study Chair — University of Alabama at Birmingham; Alexander H Paterson, MD, FRCP, Study Chair — Tom Baker Cancer Centre - Calgary; Elizabeth C. Dees, MD, Study Chair — UNC Lineberger Comprehensive Cancer Center; Mark J. Clemons, MD, Study Chair — Toronto Sunnybrook Regional Cancer Centre

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716
- [Derived] Kizub DA, Miao J, Schubert MM, Paterson AHG, Clemons M, Dees EC, Ingle JN, Falkson CI, Barlow WE, Hortobagyi GN, Gralow JR. Risk factors for bisphosphonate-associated osteonecrosis of the jaw in the prospective randomized trial of adjuvant bisphosphonates for early-stage breast cancer (SWOG 0307). Support Care Cancer. 2021 May;29(5):2509-2517. doi: 10.1007/s00520-020-05748-8. Epub 2020 Sep 15. PMID 32929540
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I Zoledronate: Patients receive zoledronate IV over 15 minutes once a month for 6 months and then once every 3 months for 2.5 years.
  zoledronic acid: Given IV
- Arm II Clodronate: Patients receive oral clodronate once daily for 35 months.
  clodronate disodium: Given orally
- Arm III Ibandronate: Patients receive oral ibandronate once daily for 35 months.
  ibandronate sodium: Given orally
Period: Overall Study
Arm/Group | Arm I Zoledronate | Arm II Clodronate | Arm III Ibandronate
Started | 2262 | 2268 | 1567
Completed | 1433 | 1295 | 955
Not Completed | 829 | 973 | 612
Not completed — Adverse Event | 228 | 387 | 273
Not completed — Death | 8 | 6 | 5
Not completed — Withdrawal by Subject | 318 | 310 | 172
Not completed — Other-non protocol specified | 142 | 129 | 77
Not completed — Data not reported | 6 | 10 | 1
Not completed — Progression | 127 | 131 | 84

BASELINE CHARACTERISTICS:
Population: Only eligible patients are included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I Zoledronate | Arm II Clodronate | Arm III Ibandronate | Total
Number analyzed (Participants) | 2231 | 2235 | 1552 | 6018
Age, Continuous [Median (Full Range); unit: years] | 53.0 [24.8 to 85.7] | 52.6 [21.2 to 86.1] | 52.7 [26.1 to 85.8] | 52.7 [21.2 to 86.1]
Age, Customized [Count of Participants; unit: Participants]
  Age, Categorized: Age < 55 | 1270 | 1304 | 894 | 3468
  Age, Categorized: Age >= 55 | 961 | 931 | 658 | 2550
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2231 | 2235 | 1552 | 6018
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 | 8 | 4 | 24
  Asian | 70 | 90 | 57 | 217
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 3 | 7
  Black or African American | 129 | 118 | 85 | 332
  White | 1975 | 1976 | 1374 | 5325
  More than one race | 12 | 5 | 2 | 19
  Unknown or Not Reported | 31 | 36 | 27 | 94
Nodal Status [Count of Participants; unit: Participants]
  Negative | 1089 | 1152 | 784 | 3025
  1~3 | 722 | 685 | 489 | 1896
  >=4 | 404 | 385 | 267 | 1056
ER/PR [Count of Participants; unit: Participants]
  Negative (ER-, PR-) | 480 | 487 | 319 | 1286
  Positive (ER+ or PR+) | 1747 | 1747 | 1231 | 4725
HER2 status [Count of Participants; unit: Participants]
  HER2 negative | 1787 | 1786 | 1247 | 4820
  HER2 positive/equivocal | 418 | 427 | 288 | 1133
Breast disease subtype [Count of Participants; unit: Participants]
  ER+ or PR+, HER2- | 1437 | 1419 | 1015 | 3871
  ER+ or PR+, HER2+ | 292 | 312 | 205 | 809
  ER/PR-, HER2- (triple neg) | 350 | 367 | 232 | 949
  ER/PR-, HER2+ (triple neg) | 126 | 115 | 83 | 324
Stage [Count of Participants; unit: Participants] — Staging criterial is per AJCC 6th Edition, 2002. Higher staging means worse disease.
  Participants
    Stage I | 721 | 770 | 509 | 2000
    Stage II | 992 | 954 | 694 | 2640
    Stage III | 472 | 460 | 304 | 1236
Chemotherapy [Count of Participants; unit: Participants]
  Not given or planned | 446 | 454 | 319 | 1219
  Given or planned | 1779 | 1778 | 1232 | 4789
Hormonal Therapy [Count of Participants; unit: Participants]
  Not given or planned | 542 | 535 | 367 | 1444
  Given or planned | 1670 | 1686 | 1170 | 4526

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival
Description: Time from date of registration to date of first observation of recurrence or death due to any cause. Patients last known to be alive who have not experienced recurrence of disease are censored at their last contact date. The outcome for the disease-free survival will be presented as 5 year survival rate.
Time Frame: Disease assessments are completed every 6 months for 5 years then annually for 5 years or until death or recurrence
Population: Only eligible patients will be included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of analyzed participants
Arm/Group | Arm I Zoledronate | Arm II Clodronate | Arm III Ibandronate
Number analyzed (Participants) | 2231 | 2235 | 1552
percentage of analyzed participants | 88 [87 to 90] | 88 [86 to 89] | 87 [86 to 89]
Statistical Analysis 1: Comparison: Arm I Zoledronate vs Arm II Clodronate vs Arm III Ibandronate; Test type: Other; p = 0.49, Log Rank
Statistical Analysis 2: Comparison: Arm I Zoledronate vs Arm II Clodronate; Test type: Superiority; p = 0.24, Regression, Cox; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.94 to 1.26]
Statistical Analysis 3: Comparison: Arm I Zoledronate vs Arm III Ibandronate; Test type: Superiority; p = 0.50, Regression, Cox; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.90 to 1.24]

2. Secondary Outcome: Overall Survival
Description: Time from date of registration to date of death due to any cause. Patients last known to be alive are censored at their last contact date. The outcome for overall survival will be presented as 5 year overall survival rate.
Time Frame: follow up completed every 6 months for 5 years and then annually for 5 years or until death
Population: Only eligible patients will be included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of analyzable patients
Arm/Group | Arm I Zoledronate | Arm II Clodronate | Arm III Ibandronate
Number analyzed (Participants) | 2231 | 2235 | 1552
percentage of analyzable patients | 93 [91 to 94] | 92 [91 to 94] | 93 [92 to 94]
Statistical Analysis 1: Comparison: Arm I Zoledronate vs Arm II Clodronate vs Arm III Ibandronate; Test type: Other; p = 0.50, Log Rank

3. Secondary Outcome: Distributions of Sites of First Recurrence on the Three Arms.
Description: All sites of invasive disease documented within 30 days of first documentation of invasive recurrence.
Time Frame: Disease assessments are completed every 6 months for 5 years then annually for 5 years or until death or recurrence
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I Zoledronate | Arm II Clodronate | Arm III Ibandronate
Number analyzed (Participants) | 2231 | 2235 | 1552
Participants
  Local/Regional only | 41 | 55 | 36
  Contralateral only | 17 | 18 | 17
  Distant recurrence | 218 | 207 | 146
  Unknown location of recurrence | 10 | 15 | 10
  Bone as 1st site of distant recurrence | 110 | 108 | 82
  Bone only | 62 | 48 | 44
  Bone and nodes only | 2 | 2 | 2
  Bone and other distant sites (beside nodes) | 46 | 58 | 36
  Liver/lung/other visceral without bone recurrence | 57 | 67 | 40
  Brain/other CNS (+/- any other site) | 31 | 24 | 22
Statistical Analysis 1: Comparison: Arm I Zoledronate vs Arm II Clodronate vs Arm III Ibandronate; Statistical analysis for recurrence to bone; Test type: Other; p = 0.93, Log Rank

4. Secondary Outcome: Number of Patients With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Adverse Events (AEs) are reported by CTCAE Version 4.0. Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Toxicity assessment is repeated every 2 months for the first 6 months, then every 3 months until 3 years or end of treatment.
Population: Patients who received at least one dose of protocol treatment.
Measure: Number; unit: Participants
Groups:
- Arm I Zoledronic Acid: Patients receive zoledronate IV over 15 minutes once a month for 6 months and then once every 3 months for 2.5 years.
  zoledronic acid: Given IV
- Arm III Ibandronate: Arm III Ibandronate
  Patients receive oral ibandronate once daily for 35 months.
  ibandronate sodium: Given orally
Arm/Group | Arm I Zoledronic Acid | Arm II Clodronate | Arm III Ibandronate
Number analyzed (Participants) | 2113 | 2169 | 1518
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 1 | 3 | 1
  AST, SGOT | 1 | 5 | 3
  Alkaline phosphatase | 0 | 1 | 0
  Allergic reaction/hypersensitivity | 2 | 1 | 1
  Anorexia | 0 | 1 | 0
  Arthritis (non-septic) | 5 | 2 | 2
  Auditory/Ear-Other (Specify) | 1 | 0 | 0
  Bilirubin (hyperbilirubinemia) | 0 | 1 | 1
  Blood/Bone Marrow-Other (Specify) | 0 | 0 | 1
  CNS cerebrovascular ischemia | 0 | 1 | 0
  Calcium, serum-low (hypocalcemia) | 3 | 2 | 1
  Cardiac General-Other (Specify) | 0 | 0 | 1
  Confusion | 0 | 1 | 0
  Constipation | 0 | 1 | 1
  Creatinine | 2 | 1 | 4
  Dehydration | 1 | 2 | 0
  Dental: periodontal disease | 2 | 0 | 0
  Dental: teeth | 0 | 1 | 0
  Diarrhea | 2 | 11 | 5
  Distention/bloating, abdominal | 0 | 1 | 0
  Dizziness | 1 | 3 | 0
  Dysphagia (difficulty swallowing) | 0 | 1 | 1
  Dyspnea (shortness of breath) | 3 | 2 | 3
  Edema: limb | 1 | 1 | 4
  Endocrine-Other (Specify) | 0 | 1 | 0
  Esophagitis | 0 | 2 | 5
  Extremity-upper (function) | 0 | 0 | 1
  Fatigue (asthenia, lethargy, malaise) | 11 | 10 | 7
  Febrile neutropenia | 1 | 1 | 0
  Fever in absence of neutropenia, ANC lt1.0x10e9/L | 1 | 1 | 0
  Flu-like syndrome | 3 | 0 | 0
  Fracture | 0 | 3 | 1
  Gastritis (including bile reflux gastritis) | 0 | 1 | 1
  Glucose, serum-high (hyperglycemia) | 0 | 2 | 0
  Heartburn/dyspepsia | 2 | 22 | 22
  Hemoglobin | 3 | 2 | 1
  Hemorrhage, GI - Rectum | 0 | 1 | 0
  Hemorrhage, GI - Stomach | 0 | 0 | 1
  Hot flashes/flushes | 3 | 5 | 4
  Hypertension | 2 | 2 | 1
  Hypotension | 0 | 1 | 0
  INR (of prothrombin time) | 0 | 1 | 0
  Incontinence, urinary | 1 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Skin | 1 | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Soft tissue | 1 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Bone | 1 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Bronchus | 0 | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Dental | 0 | 1 | 1
  Infection with unknown ANC - Appendix | 0 | 0 | 1
  Infection with unknown ANC - Liver | 1 | 0 | 0
  Infection with unknown ANC - Skin (cellulitis) | 0 | 1 | 0
  Insomnia | 1 | 3 | 0
  Irregular menses (change from baseline) | 2 | 0 | 0
  Irritability (children lt3 years of age) | 0 | 1 | 0
  Joint-function | 0 | 0 | 1
  Left ventricular systolic dysfunction | 0 | 0 | 1
  Leukocytes (total WBC) | 2 | 1 | 0
  Lymphopenia | 2 | 3 | 0
  Magnesium, serum-high (hypermagnesemia) | 1 | 2 | 0
  Magnesium, serum-low (hypomagnesemia) | 1 | 0 | 0
  Masculinization of female | 0 | 0 | 1
  Memory impairment | 1 | 0 | 0
  Metabolic/Laboratory-Other (Specify) | 0 | 1 | 0
  Mood alteration - anxiety | 0 | 0 | 1
  Mood alteration - depression | 1 | 1 | 1
  Mood alteration - euphoria | 0 | 1 | 0
  Mucositis/stomatitis (clinical exam) - Oral cavity | 1 | 0 | 0
  Muscle weakness, not d/t neuropathy - Extrem-lower | 0 | 1 | 0
  Muscle weakness, not d/t neuropathy - Extrem-upper | 0 | 1 | 0
  Muscle weakness, not d/t neuropathy - body/general | 0 | 1 | 0
  Nausea | 3 | 5 | 2
  Neuropathy: motor | 0 | 0 | 1
  Neuropathy: sensory | 0 | 6 | 4
  Neutrophils/granulocytes (ANC/AGC) | 6 | 5 | 0
  Obesity | 1 | 1 | 0
  Opportunistic inf associated w/gt=Gr 2 lymphopenia | 1 | 0 | 0
  Osteonecrosis (avascular necrosis) | 6 | 1 | 3
  Pain - Abdomen NOS | 0 | 1 | 1
  Pain - Back | 3 | 2 | 6
  Pain - Bone | 47 | 19 | 19
  Pain - Chest wall | 0 | 1 | 0
  Pain - Chest/thorax NOS | 0 | 0 | 2
  Pain - Extremity-limb | 4 | 3 | 4
  Pain - Head/headache | 8 | 3 | 1
  Pain - Joint | 39 | 35 | 42
  Pain - Muscle | 23 | 5 | 16
  Pain - Neck | 1 | 0 | 1
  Pain - Neuralgia/peripheral nerve | 1 | 0 | 0
  Pain - Oral cavity | 0 | 0 | 1
  Pain - Pain NOS | 1 | 0 | 0
  Pain - Stomach | 1 | 1 | 1
  Pain - Throat/pharynx/larynx | 0 | 0 | 1
  Pain - Vagina | 0 | 0 | 1
  Pain-Other (Specify) | 4 | 4 | 0
  Pancreatitis | 0 | 1 | 0
  Perforation, GI - Duodenum | 0 | 1 | 0
  Phosphate, serum-low (hypophosphatemia) | 19 | 6 | 8
  Platelets | 1 | 0 | 0
  Potassium, serum-high (hyperkalemia) | 0 | 0 | 1
  Potassium, serum-low (hypokalemia) | 1 | 5 | 1
  Proteinuria | 0 | 0 | 1
  Pruritus/itching | 0 | 1 | 0
  Rash/desquamation | 0 | 3 | 2
  Renal failure | 2 | 2 | 5
  Renal/Genitourinary-Other (Specify) | 0 | 0 | 3
  Retinal detachment | 1 | 0 | 0
  Rigors/chills | 1 | 0 | 0
  Secondary Malignancy-poss rel to cancer Tx | 0 | 1 | 0
  Sexual/Reproductive Function-Other (Specify) | 1 | 0 | 1
  Sodium, serum-low (hyponatremia) | 0 | 1 | 0
  Soft tissue necrosis - Head | 0 | 0 | 1
  Syncope (fainting) | 2 | 0 | 0
  Thrombosis/embolism (vascular access-related) | 1 | 1 | 0
  Thrombosis/thrombus/embolism | 0 | 0 | 1
  Tinnitus | 1 | 0 | 0
  Urticaria (hives, welts, wheals) | 1 | 2 | 1
  Vomiting | 1 | 1 | 1
  Weight gain | 0 | 1 | 0
  Weight loss | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: Toxicity assessment is repeated every 2 months for the first 6 months, then every 3 months until 3 years or end of treatment.
Description: For Adverse Event assessment, we include patients who are eligible and evaluable for adverse events (e.g., received at least one dose of protocol treatment) in the analysis. For all-cause mortality, we include all eligible patients in the analysis.
Arm/Group | Arm I Zoledronic Acid | Arm II Clodronate | Arm III Ibandronate
All-Cause Mortality (participants affected / at risk) | 238/2231 | 263/2235 | 182/1552
Serious Adverse Events (participants affected / at risk) | 21/2125 | 190/2186 | 141/1530
Other Adverse Events (participants affected / at risk) | 1854/2125 | 1942/2186 | 1366/1530
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I Zoledronic Acid (N=2125) | Arm II Clodronate (N=2186) | Arm III Ibandronate (N=1530)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 6
Hemoglobin (Blood and lymphatic system disorders) | 0 | 3 | 2
Cardiac General-Other (Cardiac disorders) | 0 | 2 | 2
Cardiac-ischemia/infarction (Cardiac disorders) | 1 | 1 | 4
Conduction abnorm/AV block - Sick sinus syndrome (Cardiac disorders) | 0 | 1 | 0
Left ventricular diastolic dysfunction (Cardiac disorders) | 0 | 3 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1 | 4
Pain - Cardiac/heart (Cardiac disorders) | 0 | 3 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (non-malignant) (Cardiac disorders) | 0 | 0 | 1
SVT and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 0 | 4 | 1
SVT and nodal arrhythmia - Atrial tachycardia/PAT (Cardiac disorders) | 0 | 1 | 0
SVT and nodal arrhythmia - SVT tachycardia (Cardiac disorders) | 0 | 2 | 0
SVT and nodal arrhythmia - Sinus bradycardia (Cardiac disorders) | 0 | 1 | 1
SVT and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Valvular heart disease (Cardiac disorders) | 0 | 0 | 1
Ventricular arrhythmia - PVCs (Cardiac disorders) | 0 | 0 | 1
Ventricular arrhythmia - Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 1
Endocrine-Other (Endocrine disorders) | 0 | 2 | 0
Ocular/Visual-Other (Eye disorders) | 0 | 0 | 1
Vision-blurred vision (Eye disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2
Dental: periodontal disease (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 4 | 2
Distention/bloating, abdominal (Gastrointestinal disorders) | 0 | 1 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 1
Fistula, GI - Colon/cecum/appendix (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal-Other (Gastrointestinal disorders) | 0 | 0 | 1
Hemorrhage, GI - Cecum/appendix (Gastrointestinal disorders) | 0 | 1 | 0
Hemorrhage, GI - Esophagus (Gastrointestinal disorders) | 0 | 1 | 0
Hemorrhage, GI - Stomach (Gastrointestinal disorders) | 0 | 0 | 1
Hemorrhage, GI - Varices (rectal) (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 5
Obstruction, GI - Cecum (Gastrointestinal disorders) | 0 | 1 | 0
Obstruction, GI - Small bowel NOS (Gastrointestinal disorders) | 0 | 5 | 0
Obstruction, GI - Stomach (Gastrointestinal disorders) | 0 | 0 | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 0 | 10 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 3 | 2
Perforation, GI - Duodenum (Gastrointestinal disorders) | 0 | 1 | 0
Ulcer, GI - Stomach (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 3
Death not associated with CTCAE term - Death NOS (General disorders) | 0 | 1 | 1
Edema: head and neck (General disorders) | 0 | 1 | 0
Edema: limb (General disorders) | 0 | 1 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 | 4 | 0
Pain - Chest/thorax NOS (General disorders) | 0 | 0 | 3
Pain - Pain NOS (General disorders) | 0 | 1 | 0
Pain-Other (General disorders) | 0 | 1 | 0
Sudden death (General disorders) | 1 | 1 | 0
Syndromes-Other (General disorders) | 1 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 4 | 7
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 0 | 0 | 1
Pain - Liver (Hepatobiliary disorders) | 0 | 1 | 0
Allergic reaction/hypersensitivity (Immune system disorders) | 0 | 4 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Blood (Infections and infestations) | 0 | 3 | 1
Inf (clin/microbio) w/Gr 3-4 neuts - Catheter-rel (Infections and infestations) | 0 | 1 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Sinus (Infections and infestations) | 0 | 1 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Skin (Infections and infestations) | 1 | 0 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Blood (Infections and infestations) | 0 | 2 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Bronchus (Infections and infestations) | 0 | 1 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Catheter (Infections and infestations) | 0 | 2 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Colon (Infections and infestations) | 0 | 2 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Kidney (Infections and infestations) | 0 | 0 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 0 | 4 | 3
Inf w/normal ANC or Gr 1-2 neutrophils - Lymphatic (Infections and infestations) | 0 | 1 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Skin (Infections and infestations) | 0 | 16 | 12
Inf w/normal ANC or Gr 1-2 neutrophils - Soft tiss (Infections and infestations) | 0 | 1 | 2
Inf w/normal ANC or Gr 1-2 neutrophils - Wound (Infections and infestations) | 0 | 2 | 0
Inf w/normal ANC or Gr 1-2 neutrophils-Foreign bod (Infections and infestations) | 0 | 0 | 2
Infection with normal ANC or Grade 1 or 2 neutroph (Infections and infestations) | 0 | 1 | 1
Infection with unknown ANC - Appendix (Infections and infestations) | 0 | 1 | 1
Infection with unknown ANC - Blood (Infections and infestations) | 0 | 0 | 1
Infection with unknown ANC - Bronchus (Infections and infestations) | 0 | 1 | 0
Infection with unknown ANC - Catheter-related (Infections and infestations) | 0 | 0 | 1
Infection with unknown ANC - Duodenum (Infections and infestations) | 0 | 0 | 1
Infection with unknown ANC - Foreign body (e.g., g (Infections and infestations) | 0 | 1 | 1
Infection with unknown ANC - Heart (endocarditis) (Infections and infestations) | 0 | 0 | 1
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 0 | 2 | 3
Infection with unknown ANC - Skin (cellulitis) (Infections and infestations) | 0 | 10 | 3
Infection with unknown ANC - Soft tissue NOS (Infections and infestations) | 0 | 2 | 0
Infection with unknown ANC - Upper airway NOS (Infections and infestations) | 0 | 0 | 1
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 0 | 0 | 1
Infection with unknown ANC - Wound (Infections and infestations) | 0 | 7 | 1
Infection-Other (Infections and infestations) | 0 | 2 | 3
Fracture (Injury, poisoning and procedural complications) | 0 | 11 | 10
Intra-operative Injury-Other (Injury, poisoning and procedural complications) | 0 | 1 | 0
Intra-operative injury - Ovary (Injury, poisoning and procedural complications) | 0 | 0 | 1
Leak (including anastomotic), GI - Leak NOS (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rash: dermatitis associated w/radiation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 0 | 1 | 1
Vessel injury-artery - Carotid (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound complication, non-infectious (Injury, poisoning and procedural complications) | 0 | 0 | 2
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 0 | 5 | 1
AST, SGOT (Investigations) | 0 | 4 | 2
Alkaline phosphatase (Investigations) | 0 | 1 | 0
Bilirubin (hyperbilirubinemia) (Investigations) | 0 | 1 | 0
Creatinine (Investigations) | 0 | 1 | 1
Leukocytes (total WBC) (Investigations) | 0 | 3 | 2
Lymphopenia (Investigations) | 0 | 1 | 0
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 0 | 5 | 3
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 0 | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 8 | 4
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 0 | 2 | 0
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 0 | 3 | 0
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 | 1 | 0
Pancreatic endocrine: glucose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 1
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 | 2 | 2
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 0 | 1 | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 | 3 | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 | 3 | 0
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal/Soft Tissue-Other (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 13 | 5 | 5
Pain - Back (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Pain - Bone (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain - Joint (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Pain - Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Secondary Malignancy-poss rel to cancer Tx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1
Ataxia (incoordination) (Nervous system disorders) | 0 | 1 | 1
CNS cerebrovascular ischemia (Nervous system disorders) | 0 | 4 | 4
Cognitive disturbance (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 5 | 1
Hemorrhage, CNS (Nervous system disorders) | 0 | 1 | 0
Neurology-Other (Nervous system disorders) | 0 | 1 | 2
Neuropathy: CN VII Motor-face; Sensory-taste (Nervous system disorders) | 0 | 0 | 1
Neuropathy: motor (Nervous system disorders) | 0 | 1 | 2
Neuropathy: sensory (Nervous system disorders) | 0 | 2 | 1
Ocular/Visual-Other (Nervous system disorders) | 0 | 0 | 1
Pain - Head/headache (Nervous system disorders) | 0 | 7 | 0
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1
Syncope (fainting) (Nervous system disorders) | 0 | 3 | 5
Vasovagal episode (Nervous system disorders) | 0 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 2 | 1
Mood alteration - depression (Psychiatric disorders) | 0 | 3 | 1
Personality/behavioral (Psychiatric disorders) | 0 | 1 | 0
Cystitis (Renal and urinary disorders) | 0 | 0 | 1
Glomerular filtration rate (Renal and urinary disorders) | 0 | 1 | 0
Hemorrhage, GU - Ureter (Renal and urinary disorders) | 0 | 0 | 1
Hemorrhage, GU - Urinary NOS (Renal and urinary disorders) | 0 | 0 | 1
Obstruction, GU - Ureter (Renal and urinary disorders) | 0 | 1 | 1
Pain - Bladder (Renal and urinary disorders) | 0 | 0 | 1
Pain - Kidney (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 2 | 0
Renal/Genitourinary-Other (Renal and urinary disorders) | 0 | 2 | 2
Hemorrhage, GU - Uterus (Reproductive system and breast disorders) | 0 | 1 | 0
Sexual/Reproductive Function-Other (Reproductive system and breast disorders) | 1 | 0 | 4
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 10 | 9
Hemorrhage, pulmonary/upper respiratory - Larynx (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hematoma (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 2 | 0
Phlebitis (including superficial thrombosis) (Vascular disorders) | 0 | 0 | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 9 | 10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I Zoledronic Acid (N=2125) | Arm II Clodronate (N=2186) | Arm III Ibandronate (N=1530)
Hemoglobin (Blood and lymphatic system disorders) | 376 | 326 | 251
Constipation (Gastrointestinal disorders) | 230 | 259 | 180
Diarrhea (Gastrointestinal disorders) | 288 | 447 | 223
Heartburn/dyspepsia (Gastrointestinal disorders) | 138 | 332 | 280
Nausea (Gastrointestinal disorders) | 454 | 555 | 307
Pain - Abdomen NOS (Gastrointestinal disorders) | 133 | 146 | 100
Vomiting (Gastrointestinal disorders) | 158 | 243 | 123
Edema: limb (General disorders) | 243 | 212 | 163
Fatigue (asthenia, lethargy, malaise) (General disorders) | 851 | 749 | 560
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 261 | 82 | 70
Flu-like syndrome (General disorders) | 108 | 24 | 18
Pain-Other (General disorders) | 185 | 149 | 122
Rigors/chills (General disorders) | 109 | 27 | 18
Rash: dermatitis associated w/radiation (Injury, poisoning and procedural complications) | 108 | 100 | 70
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 290 | 540 | 170
AST, SGOT (Investigations) | 308 | 581 | 190
Alkaline phosphatase (Investigations) | 114 | 166 | 77
Creatinine (Investigations) | 205 | 230 | 127
Leukocytes (total WBC) (Investigations) | 366 | 370 | 205
Lymphopenia (Investigations) | 209 | 181 | 125
Metabolic/Laboratory-Other (Investigations) | 120 | 132 | 67
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 160 | 213 | 100
Platelets (Investigations) | 118 | 140 | 51
Weight gain (Investigations) | 124 | 137 | 81
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 109 | 97 | 61
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 196 | 162 | 111
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 484 | 429 | 283
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 119 | 84 | 58
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 120 | 88 | 82
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 148 | 87 | 80
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 172 | 189 | 88
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 114 | 106 | 78
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 206 | 197 | 143
Pain - Back (Musculoskeletal and connective tissue disorders) | 295 | 253 | 213
Pain - Bone (Musculoskeletal and connective tissue disorders) | 614 | 390 | 303
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 260 | 231 | 173
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1071 | 968 | 756
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 488 | 339 | 294
Dizziness (Nervous system disorders) | 196 | 157 | 134
Neuropathy: sensory (Nervous system disorders) | 464 | 447 | 311
Pain - Head/headache (Nervous system disorders) | 310 | 270 | 205
Insomnia (Psychiatric disorders) | 345 | 310 | 204
Mood alteration - anxiety (Psychiatric disorders) | 178 | 159 | 106
Mood alteration - depression (Psychiatric disorders) | 236 | 227 | 151
Pain - Breast (Reproductive system and breast disorders) | 129 | 144 | 102
Vaginal dryness (Reproductive system and breast disorders) | 128 | 137 | 90
Cough (Respiratory, thoracic and mediastinal disorders) | 216 | 216 | 143
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 185 | 133 | 116
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 138 | 120 | 90
Rash/desquamation (Skin and subcutaneous tissue disorders) | 306 | 307 | 194
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 97 | 97 | 79
Hot flashes/flushes (Vascular disorders) | 795 | 808 | 579
Hypertension (Vascular disorders) | 94 | 127 | 60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2014-12-19): https://cdn.clinicaltrials.gov/large-docs/05/NCT00127205/Prot_SAP_ICF_000.pdf